CLINICAL TRIAL: NCT02904395
Title: Feasability and Interest of Screening for Infantile Pompe's Diseases at Birth
Acronym: DEPIPOMP1
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier de Cayenne (Other)
Responsible Party: Sponsor
Other Study IDs: DEPIPOMP1
Record Dates: First submitted 2016-09-06; First posted 2016-09-19 (Estimated); Last update posted 2016-09-19 (Estimated); Status verified 2016-09

CONDITIONS: Pompe's Disease
MeSH Terms: conditions — Glycogen Storage Disease Type II

STUDY DESIGN:
Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — filter paper with blood to look for enzyme activity and if enzyme activity low, PCR looking for the signature mutations for infantile Pompe's Disease
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: observational (no intervention)

SUMMARY:
Given the 100 fold increase of the incidence of Pompe's disease in Western French Guiana, the objective of the present study is to implement systematic screening in newborns in French Guiana in order to start treatment before the muscular and cardiac symptoms appear.

ELIGIBILITY:
Inclusion Criteria:

* newborn

Exclusion Criteria:

* parent refusal

Max Age: 2 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: newborns
Sampling Method: Non-Probability Sample
Enrollment: 3413 (Actual)
Dates: Start 2014-04; Primary Completion 2014-04 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
acid maltase activity | At birth
  The acid maltase enzyme activity is evaluated just after birth. If it is abnormal then PCR allows to identify signature mutations.
Signature mutation for pompe's disease | At birth
  The acid maltase enzyme activity is evaluated just after birth. If it is abnormal then PCR allows to identify signature mutations.

IPD SHARING:
Plan to Share IPD: No